CLINICAL TRIAL: NCT01746888
Title: Expanding Antimicrobial Stewardship
Status: Completed | Type: Observational
Sponsor: Jeffrey Caterino (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Caterino, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2011H0165
Record Dates: First submitted 2012-10-23; First posted 2012-12-11 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Older Adults: Adults 65 years and older who present to the Emergency Department.

SUMMARY:
Gold standard diagnostic criteria for diagnosing acute infection in older adult patients in the Emergency Department do not currently exist. These patients often have atypical presentations which can complicate diagnosis and treatment. The development of an antimicrobial stewardship program for Emergency Department older adult patients can ultimately improve the accuracy of diagnosis and correct antimicrobial prescribing. This research study involves data collection from enrolled subjects and treating physicians. The data will be collected using a patient interview which will be answered directly by the patient or caregiver. Additional surveys will be administered to the Emergency Department treating physician and subsequent physician. Additional data will be abstracted from the Emergency Department chart and from additional charts that often accompanies the patient to the Emergency Department. A physician adjudication process will occur if there is disagreement in diagnosis between the treating Emergency Department physician and succeeding physician.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age

Exclusion Criteria:

* Patient incarcerated
* Chief complaint of suicidal or homicidal ideation
* Patient primarily evaluated by the trauma team

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Adults 65 years of age and older who present to the Emergency Department.
Sampling Method: Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Presence of infection while in the Emergency Department | participants will be followed for the duration of hospital stay, an expected average of 4 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Caterino, MD, MPH, Principal Investigator — Ohio State University
Locations (1):
- Wexner Medical Center at The Ohio State University, Columbus, Ohio, United States